CLINICAL TRIAL: NCT02216526
Title: A Prevalence and Multi-center Randomized Parallel-group Pragmatic Trial to Compare the Effectiveness of Standardized Skin Care Regimens on Skin Health in Nursing Home Residents
Brief Title: Skin Health and Effectiveness of Standardized Skin Care Regimens in Nursing Home Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PD Dr. Jan Kottner (Other)
Responsible Party: Sponsor-Investigator, PD Dr. Jan Kottner, Scientific Director Clinical Research Center for Hair and Skin Science, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRC-SP-A-15
Record Dates: First submitted 2014-08-11; First posted 2014-08-15 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Xerosis Cutis
Keywords: Skin health; Nursing; Long-term care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cetaphil® Restoraderm (Experimental): Cetaphil® Restoraderm Body Wash, once daily for 8 weeks and Cetaphil® Restoraderm Body Moisturizer, twice daily for 8 weeks
  Interventions: Other: Cetaphil® Restoraderm
- Excipial (Experimental): Excipial Kids Body Wash, once daily for 8 weeks and Excipial U Lipolotio (4% urea), twice daily for 8 weeks
  Interventions: Other: Excipial
- Standard skin care (No Intervention): Usual skin care routine of the nursing home resident

INTERVENTIONS:
Other: Cetaphil® Restoraderm
  Arms: Cetaphil® Restoraderm
Other: Excipial
  Arms: Excipial

SUMMARY:
Residents of institutional long-term care facilities are at high risk for developing skin and tissue diseases, e.g. xerosis cutis (including pruritus), infections (e.g., tinea pedis, candidiasis), chronic wounds or neoplastic changes (e.g. actinic keratosis, malignant melanoma) but there are few epidemiological figures about the actual frequencies of these conditions in nursing homes. Therefore, in the first part of this study we aim at measuring key dermatological conditions and associated health and functional status, and the skin care practice of aged nursing home residents ("prevalence study").

Basic skin care interventions are believed to reduce skin dryness and to enhance skin health. Thus, the second aim of this study is to investigate the effectiveness of two structured skin care regimens compared to the routine standard skin care on skin health in nursing home residents ("intervention study").

The study will be conducted in a random sample of seven out of approximately 300 institutional long term care facilities of the federal state of Berlin.

ELIGIBILITY:
Inclusion Criteria:

"Prevalence study"

* Living in the nursing home at the time of data collection;
* Being 65+ years;
* Written informed consent (or by legal representative);

Additional inclusion criteria for the "intervention study"

* Overall dry skin score (ODS) of 2 to 4 at the right and left leg;
* Willingness and ability to fulfil the study requirements.

Exclusion Criteria:

"Prevalence study"

* Residents at the end of life (dying persons).

Additional exclusion criteria for the "intervention study"

* Any dermatological condition or skin affection, e.g. acute weeping, excoriated or inflammatory dermatitis, or skin treatment which may interfere with the study assessments at the discretion of the investigator;
* Any unstable acute or chronic pathology or condition that may interfere with the study conduct at the discretion of the investigator;
* Any use of topical drugs on the investigational areas two weeks prior to inclusion;
* Systemic application of corticosteroids, antihistamine or other anti-inflammatory drugs;
* Known allergy or intolerance to any ingredient of the study products, e.g. urea.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Blume-Peytavi, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gabriel S, Hahnel E, Blume-Peytavi U, Kottner J. Prevalence and associated factors of intertrigo in aged nursing home residents: a multi-center cross-sectional prevalence study. BMC Geriatr. 2019 Apr 15;19(1):105. doi: 10.1186/s12877-019-1100-8. PMID 30987588
- [Derived] Hahnel E, Blume-Peytavi U, Trojahn C, Kottner J. Associations between skin barrier characteristics, skin conditions and health of aged nursing home residents: a multi-center prevalence and correlational study. BMC Geriatr. 2017 Nov 13;17(1):263. doi: 10.1186/s12877-017-0655-5. PMID 29132305
- [Derived] Hahnel E, Blume-Peytavi U, Trojahn C, Dobos G, Jahnke I, Kanti V, Richter C, Lichterfeld-Kottner A, Garcia Bartels N, Kottner J. Prevalence and associated factors of skin diseases in aged nursing home residents: a multicentre prevalence study. BMJ Open. 2017 Sep 24;7(9):e018283. doi: 10.1136/bmjopen-2017-018283. PMID 28947467
- [Derived] Hahnel E, Blume-Peytavi U, Trojahn C, Dobos G, Stroux A, Garcia Bartels N, Jahnke I, Lichterfeld-Kottner A, Neels-Herzmann H, Klasen A, Kottner J. The effectiveness of standardized skin care regimens on skin dryness in nursing home residents: A randomized controlled parallel-group pragmatic trial. Int J Nurs Stud. 2017 May;70:1-10. doi: 10.1016/j.ijnurstu.2017.02.006. Epub 2017 Feb 7. PMID 28214613
- [Derived] Kottner J, Hahnel E, Trojahn C, Stroux A, Dobos G, Lichterfeld A, Richter C, Blume-Peytavi U. A multi-center prevalence study and randomized controlled parallel-group pragmatic trial to compare the effectiveness of standardized skin care regimens on skin health in nursing home residents: a study protocol. Int J Nurs Stud. 2015 Feb;52(2):598-604. doi: 10.1016/j.ijnurstu.2014.11.007. Epub 2014 Nov 15. PMID 25443420

RESULTS

PARTICIPANT FLOW:
Recruitment Details: completed, recruitment period: September 2014 to May 2015, nursing homes
Groups:
- Cetaphil® Restoraderm: Cetaphil® Restoraderm Body Wash, once daily for 8 weeks and Cetaphil® Restoraderm Body Moisturizer, twice daily for 8 weeks
  Cetaphil® Restoraderm
- Excipial: Excipial Kids Body Wash, once daily for 8 weeks and Excipial U Lipolotio (4% urea), twice daily for 8 weeks
  Excipial
Period: Overall Study
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Started | 45 | 44 | 44
Completed | 40 | 41 | 36
Not Completed | 5 | 3 | 8
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Death | 0 | 1 | 3
Not completed — Protocol Violation | 2 | 0 | 2
Not completed — Hospitalization | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care | Total
Number analyzed (Participants) | 45 | 44 | 44 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 45 | 44 | 44 | 133
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 32 | 30 | 87
  Male | 20 | 12 | 14 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 45 | 44 | 44 | 133

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Overall Dry Skin Score (ODS)
Description: Clinical assessment of the presence or severity of skin dryness using a five point rating scale at right lower leg. The Overall Dry Skin score is a clinical assessment of the presence and severity of skin dryness using a five-point scale. A score of '0' indicates no skin dryness, whereas a score of '4' indicates advanced skin roughness, large scales, inflammation and cracks.
Time Frame: Baseline; Day 56+/-4
Population: At Day 56 +/- 3 data of two participants to calculate the Change from Baseline to Day 56 +/-3 were missing. In Group I (Cetaphil) 39/40 participants were analyzed. In Group III (Standard Skin care) 35/36 participants were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 39 | 41 | 35
units on a scale | -0.9 (1.9) | -1.2 (1.1) | -0.9 (1.0)

2. Secondary Outcome: Stratum Corneum Hydration (SCH)
Description: Change in Stratum corneum hydration (SCH) at the lower leg. Instrumental skin measurements were conducted to characterize possible effects of the interventions in terms of skin function. The stratum corneum hydration was measured using the Corneometer CM 825 (Courage + Khazaka, Cologne, Germany). This measurement is based on the differences of the dielectric constant of water and other substances. With this device, only the moisture content in the stratum corneum is measured. The arbitrary units (a.u.) range from 0 to 120 where as higher readings indicate higher stratum corneum hydration.Values > 40 a.u. are often considered 'normal', whereas values < 40 a.u. are regarded as typical for dry Skin.
Time Frame: Baseline, Day 56 +/- 4
Population: At Day 56 +/- 3 data of four participants to calculate the change from Baseline to Day 56 +/-3 were missing. In Group I (Cetaphil) 39/40 participants were analyzed. In Group II (Excipial) 40/41 participants were analyzed. In Group III (Standard Skin care) 34/36 participants were analyzed.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 39 | 40 | 34
arbitrary units | 2.8 (8.9) | 1.6 (10.1) | 2.0 (8.9)

3. Secondary Outcome: Transepidermal Water Loss (TEWL)
Description: Change in Transepidermal water loss (TEWL) at the lower leg. Transepidermal water loss was measured with the Tewameter TM 300 (Courage + Khazaka, Cologne, Germany). The probe captures the constant permeation of water through the stratum corneum in gram per hour per m2. The measuring probe contains a pair of sensors that are located in different distances to the skin surface to determine temperature and relative humidity above the skin surface. The humidity gradient between both sensors is used for calculating the transepidermal water loss. Higher values indicate a higher transepidermal water loss.
Time Frame: Baseline, Day 56 +/- 4
Population: At Day 56 +/- 3 data of twelve participants to calculate the change from Baseline to Day 56 +/-3 were missing. In Group I (Cetaphil) 36/40 participants were analyzed. In Group II (Excipial) 38/41 participants were analyzed. In Group III (Standard Skin care) 31/36 participants were analyzed.
Measure: Mean (Standard Deviation); unit: g/m2/h
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 36 | 38 | 31
g/m2/h | 1.8 (11.4) | 1.4 (12.3) | 3.4 (7.0)

4. Secondary Outcome: Skin Surface pH
Description: Changes in Skin surface pH at the lower leg. Skin surface pH was measured with the Skin-pH-Meter PH 905 (Courage + Khazaka, Cologne, Germany), a planar glass electrode. The pH is a measure of acidity and alkalinity of a solution and it indicates the concentration of the hydrogen ions in an aqueous solution. Reference values of human skin have been reported to range from 4 to 6.
Time Frame: Baseline, Day 56 +/- 4
Population: At Day 56 +/- 3 data of six participants to calculate the change from Baseline to Day 56 +/-3 were missing. In Group I (Cetaphil) 39/40 participants were analyzed. In Group II (Excipial) 40/41 participants were analyzed. In Group III (Standard Skin care) 32/36 participants were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 39 | 40 | 32
units on a scale | 0.07 (0.7) | 0.3 (0.8) | 0.1 (0.7)

5. Secondary Outcome: Itch Assessment. Question 1. Hours of Itching (1 = Less Than 6 Hours/Day; 2 = 6-12 Hours/Day; 3 = 12-18 Hours/Day; 4 = 18-23hours/Day; 5 = All Day) at Baseline
Description: Self-completion of the 5-D itch scale. Having a 6-CIT score of 7 or lower was the criterion to administer the 5-D itch scale.The score of the 5-D Itch scale ranges from '5' (no pruritus) to '25' (most severe pruritus) and contains five items measuring pruritus over the past two weeks.
  A possible cognitive impairment was tested using the Six Item Cognitive Impairment Test on Day 0. It includes six simple questions, for example 'What year is it?' or 'Count backwards from 20 to 10. Scores may range from 0 (= no sign of cognitive impairment) to a maximum score of 28 (= significant cognitive impairment). Residents with sum scores > 8 were classified as 'cognitively impaired'.
Time Frame: Baseline
Population: Only participants not being cognitively impaired were able to answer the questionnaires (in total n = 32/133 at baseline).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 12 | 9 | 11
units on a scale | 1.3 (1.1) | 1.0 (0.0) | 1.0 (0.0)

6. Secondary Outcome: Number of Participants With a Pressure Ulcer at Baseline
Description: Clinical assessment of the presence of a pressure ulcer.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 45 | 44 | 44
Participants | 2 | 7 | 3

7. Secondary Outcome: Number of Participants With Incontinence Associated Dermatitis (IAD) at Baseline
Description: Clinical assessment of the presence of incontinence associated dermatitis according to the IAD-IT classification
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 45 | 44 | 44
Participants | 16 | 19 | 12

8. Secondary Outcome: Quality of Sleep. Question 1. Light Sleep (0) - Deep Sleep (10) at Baseline
Description: Self-completion of the Richards-Campbell Sleep Questionnaire (RCSQ).Sleep quality was assessed with the Pittsburgh Richard Campbell Sleep Quality Assessment. Five questions were asked regarding the sleep quality for the last night via 0-100mm visual analogue scales. The interrater reliability and the most usefulness was recently supported.
Time Frame: Baseline
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 12 | 9 | 11
units on a scale | 6.1 (3.9) | 7.1 (2.9) | 6.2 (2.9)

9. Secondary Outcome: Quality of Life Sum Score at Baseline
Description: Self-completion of the WHO-Five Well-being Index. Well-being was assessed with the WHO-Five Well-being Index. The German version of the questionnaire published by the World Health Organization in 1998 was used. Scores range from '5' (all the time) to '0' (never) for in total five items. Simple questions were asked regarding well-being in the last two weeks, e.g. 'In the last two weeks … I was happy' or '…I was relaxed'. The sum scores range from 0, indicating the lowest well-being, to 25, indicating the highest well-being. A cut-off score of < 13 is recommended. The validity and reliability of the questionnaire was recently supported.
Time Frame: Baseline
Population: Only residents being cognitively not impaired were able to answer the questionnaires (At baseline n = 32/133)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 12 | 9 | 11
units on a scale | 16.42 (4.69) | 18.33 (4.18) | 11.09 (7.37)

10. Secondary Outcome: Number of Participants With Pressure Ulcer at Day 28 +/-3
Description: Clinical assessment of the presence of pressure ulcer.
Time Frame: Day 28 +/-3
Population: After 4 weeks of the study, in total n= 13 participants were loss to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 41 | 42 | 37
Participants | 1 | 3 | 0

11. Secondary Outcome: Number of Participants With Pressure Ulcer at Day 56 +/-3
Description: Clinical assessment of the presence of a pressure ulcer.
Time Frame: Day 56 +/-3
Population: At the end of the study, in total n = 16 participants were loss to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 40 | 41 | 36
Participants | 2 | 3 | 0

12. Secondary Outcome: Number of Participants With Skin Tears at Baseline
Description: Clinical assessment of the presence of skin tears according to the STAR Classification
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 45 | 44 | 44
Participants | 2 | 1 | 5

13. Secondary Outcome: Number of Participants With Skin Tears at Day 28 +/-3
Description: Clinical assessment aof the presence of skin tears according to the STAR Classification
Time Frame: Day 28 +/-3
Population: In total n = 13 participants were loss to follow up after 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 41 | 42 | 37
Participants | 1 | 1 | 4

14. Secondary Outcome: Number of Participants With Skin Tears at Day 56 +/-3
Description: Clinical assessment aof the presence of skin tears according to the STAR Classification
Time Frame: Day 56 +/-3
Population: In total n = 16 participants were loss to follow up after eight weeks (end of the study).
Measure: Count of Participants; unit: Participants
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 40 | 41 | 36
Participants | 2 | 0 | 3

15. Secondary Outcome: Number of Participants With Incontinence Associated Dermatitis (IAD) at Day 28 +/-3
Description: Clinical assessment of the presence and/or severity of incontinence associated dermatitis according to the IAD-IT classification
Time Frame: Day 28 +/-3
Population: In total n = 13 participants were loss to follow up after 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 41 | 42 | 47
Participants | 20 | 18 | 21

16. Secondary Outcome: Number of Participants With Incontinence Associated Dermatitis (IAD) at Day 56 +/-3
Description: as for outcome 15
Time Frame: Day 56 +/-3
Population: In total n = 16 participants were loss to follow up after eight weeks (end of the study).
Measure: Count of Participants; unit: Participants
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 40 | 41 | 36
Participants | 8 | 13 | 9

17. Secondary Outcome: Quality of Life Sum Score at Day 56 +/-3
Description: as for outcome 9
Time Frame: Day 56 +/-3
Population: Only residents being cognitively not impaired were able to answer the questionnaires (in total n = 28/117 at the end of the study).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 11 | 8 | 9
units on a scale | 17.55 (5.22) | 19.00 (5.76) | 14.00 (5.52)

18. Secondary Outcome: Quality of Sleep. Question 2. Never Fall Asleep (0) - Immediately Fall Asleep (10) at Baseline
Description: as for outcome 8
Time Frame: Baseline
Population: Only residents being not cognitively impaired were able to answer the questionnaires (in total n = 32/133).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 12 | 9 | 11
units on a scale | 6.8 (3.7) | 7.2 (3.4) | 6.5 (3.2)

19. Secondary Outcome: Quality of Sleep. Question 3. Awake All Night (0) - Awake Very Little (10) at Baseline
Description: as for outcome 8
Time Frame: Baseline
Population: Only residents being not cognitively impaired were able to answer the questionnaires (in total n = 32/133 at baseline).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 12 | 9 | 11
units on a scale | 7.6 (2.6) | 8.4 (2.1) | 7.0 (2.6)

20. Secondary Outcome: Quality of Sleep. Question 4. Not Back to Sleep (0) - Back to Sleep Immediately (10) at Baseline
Description: as for outcome 8
Time Frame: Baseline
Population: Only residents being not cognitively impaired were able to answer the questionnaires (in total 32/133 at baseline).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 12 | 9 | 11
units on a scale | 7.1 (3.9) | 8.4 (2.3) | 7.8 (3.0)

21. Secondary Outcome: Quality of Sleep. Question 5. Bad Sleep (0) - Good Sleep (10) at Baseline
Description: as for outcome 8
Time Frame: Baseline
Population: Only residents not being cognitively impaired were able to answer the questionnaires (in total n = 32/133 at baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 12 | 9 | 11
units on a scale | 7.1 (2.9) | 7.5 (2.8) | 7.0 (2.9)

22. Secondary Outcome: Quality of Sleep. Question 1. Light Sleep (0) - Deep Sleep (10) at Day 56 +/-3
Description: as for outcome 8
Time Frame: Day 56 +/-3
Population: Only residents not being cognitively impaired were able to answer the questionnaires. Due to loss to follow up only n = 28/117 participants were able to answer at the end of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 11 | 8 | 9
units on a scale | 7.1 (2.9) | 7.9 (2.2) | 7.4 (2.8)

23. Secondary Outcome: Quality of Sleep. Question 2. Never Fall Asleep (0) - Immediately Fall Asleep (10) at Day 56 +/-3
Description: as for outcome 8
Time Frame: Day 56 +/-3
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 11 | 8 | 99
units on a scale | 7.9 (2.9) | 7.1 (2.8) | 8.0 (2.8)

24. Secondary Outcome: Quality of Sleep. Question 3. Awake All Night (0) - Awake Very Little (10) at Day 56 +/-3
Description: as for outcome 8
Time Frame: Day 56 +/-3
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 11 | 8 | 9
units on a scale | 6.9 (2.9) | 7.5 (2.1) | 7.1 (2.5)

25. Secondary Outcome: Quality of Sleep. Question 4. Not Back to Sleep (0) - Back to Sleep Immediately (10) at Day 56 +/-3
Description: as for outcome 8
Time Frame: Day 56 +/-3
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 11 | 8 | 9
units on a scale | 6.6 (3.4) | 9.3 (0.6) | 7.8 (3.1)

26. Secondary Outcome: Quality of Sleep. Question 5. Bad Sleep (0) - Good Sleep (10) at Day 56 +/-3
Description: as for outcome 8
Time Frame: Day 56 +/-3
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 11 | 8 | 9
units on a scale | 7.3 (3.1) | 8.1 (2.3) | 7.7 (2.8)

27. Secondary Outcome: Itch Assessment. Question 2. Itch Intensity (1 = Not Present; 2 = Mild; 3 = Moderate; 4 = Severe; 5 = Unbearable) at Baseline
Description: as for outcome 5
Time Frame: Baseline
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 12 | 9 | 11
units on a scale | 1.6 (0.7) | 2.0 (1.0) | 1.9 (0.9)

28. Secondary Outcome: Itch Assessment. Question 3. Changes in Intensity of Itch (Past Two Weeks). (1 = Completely Resolved; 2 = Much Better But Still Present; 3 = Little Bit Better, But Still Present; 4 = Unchanged, 5 = Getting Worse) at Baseline
Description: as for outcome 5
Time Frame: Baseline
Population: Only participants not being cognitively impaired were able to answer the quastionnaires (in total n = 32/133 at baseline). One value in the Excipial Group is missing for this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 12 | 8 | 11
units on a scale | 3.0 (1.5) | 4.0 (0.0) | 3.3 (1.3)

29. Secondary Outcome: Itch Assessment. Question 4. Affecting of Sleep (See Score Informations in the Outcome Measure Description) at Baseline
Description: Self-completion of the 5-D itch scale. Question 4: 1=Never affects sleep;2=Occasionally delays falling asleep;3=Frequently delays falling asleep;4=Delays falling asleep and occasionally wakes me up;5=Delays falling asleep and frequently wakes me up at night.
  Having a 6-CIT score of 7 or lower was the criterion to administer the 5-D itch scale.The score of the 5-D Itch scale ranges from '5' (no pruritus) to '25' (most severe pruritus) and contains five items measuring pruritus over the past two weeks.
  A possible cognitive impairment was tested using the Six Item Cognitive Impairment Test on Day 0. It includes six simple questions, for example 'What year is it?' or 'Count backwards from 20 to 10. Scores may range from 0 (= no sign of cognitive impairment) to a maximum score of 28 (= significant cognitive impairment). Residents with sum scores > 8 were classified as 'cognitively impaired'.
Time Frame: Baseline
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 12 | 9 | 11
units on a scale | 1.2 (0.6) | 1.2 (0.7) | 1.4 (0.5)

30. Secondary Outcome: Itch Assessment. Question 5. Affecting of Daily Activities ( 1 = Never Affects Activity; 2 = Rarely Affects Activity; 3 = Occasionally Affects Activity; 4 = Frequently Affects Activity; 5 = Always Affects Activity) at Baseline
Description: as for outcome 5
Time Frame: Baseline
Population: Only participants not being cognitively impaired were able to answer the questionnaires (in total n = 32/133 at baseline). One value in the Cetaphil Group is missing for this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 10 | 8 | 9
units on a scale | 1.1 (0.3) | 1.4 (0.7) | 1.6 (0.7)

31. Secondary Outcome: Itch Assessment. Question 1. Hours of Itching (1 = Less Than 6hours/Day; 2 = 6-12 Hours/Day; 3 = 12-18 Hours/Day; 4 = 18-23hours/Day; 5 = All Day) at Day 56 +/-3
Description: as for outcome 5
Time Frame: Day 56 +/-3
Population: Only participants not being cognitively impaired were able to answer the questionnaires. Due to a number of loss to follow up at the end of the study, n = 28/117 answer these question. In the Excipial Group one value is missing for that question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 11 | 7 | 9
units on a scale | 1.0 (0.0) | 1.1 (0.4) | 1.0 (0.0)

32. Secondary Outcome: Itch Assessment. Question 2. Itch Intensity (1 = Not Present; 2 = Mild; 3 = Moderate; 4 = Severe; 5 = Unbearable) at Day 56 +/-3
Description: as for outcome 5
Time Frame: Day 56 +/-3
Population: Only participants not being cognitively impaired were able to answer the questionnaires. Due to a number of loss to follow up at the end of the study, n = 28/117 answer these question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 11 | 8 | 9
units on a scale | 1.7 (1.0) | 1.8 (0.7) | 1.9 (0.9)

33. Secondary Outcome: Itch Assessment. Question 3. Changes in Intensity of Itch (Past Two Weeks). (1 = Completely Resolved; 2 = Much Better But Still Present; 3 = Little Bit Better, But Still Present; 4 = Unchanged, 5 = Getting Worse) at Day 56 +/-3
Description: as for outcome 5
Time Frame: Day 56 +/-3
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 11 | 8 | 9
units on a scale | 2.8 (1.8) | 2.9 (1.6) | 3.3 (1.6)

34. Secondary Outcome: Itch Assessment. Question 4. Affecting of Sleep (See Score Details in the Outcome Measure Description) at Day 56 +/-3
Description: as for outcome 29
Time Frame: Day 56 +/-3
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 11 | 8 | 9
units on a scale | 1.2 (0.4) | 1.0 (0.0) | 1.2 (0.4)

35. Secondary Outcome: Itch Assessment. Question 5. Affecting of Daily Activities ( 1 = Never Affects Activity; 2 = Rarely Affects Activity; 3 = Occasionally Affects Activity; 4 = Frequently Affects Activity; 5 = Always Affects Activity) at Day 56 +/-3
Description: as for outcome 5
Time Frame: Day 56 +/-3
Population: Only participants not being cognitively impaired were able to answer the questionnaires. Due to a number of loss to follow up at the end of the study, n = 28/117 answer these question. In the Cetaphil Group one value is missing for that question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Number analyzed (Participants) | 10 | 8 | 9
units on a scale | 1.2 (0.4) | 1.1 (0.4) | 1.3 (0.5)

ADVERSE EVENTS:
Time Frame: Undesirable effects, defined as any adverse reaction clearly linked to the normal or reasonably foreseeable use of a cosmetic product, were monitored from the time informed consent was obtained until study completion, an average of 10 weeks. All subjects experiencing undesirable effects were monitored until symptoms subsided, or until there was a satisfactory explanation for the changes observed.
Description: The intensity of the undesirable effect was described in terms of mild, moderate or severe.
Arm/Group | Cetaphil® Restoraderm | Excipial | Standard Skin Care
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 3/45 | 1/44 | 0/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetaphil® Restoraderm (N=45) | Excipial (N=44) | Standard Skin Care (N=44)
Itch and redness on arms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Intensity was mild, products were withdrawn
Erythema face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Intensity was moderate, Dose was reduced, facial application was stopped
Redness, irritation at the whole body (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Intensity was severe, Products were withdrawn
Skin dryness at the back (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Intensity was mild, products were withdrawn

LIMITATIONS AND CAVEATS:
Residents, care givers, and study personnal was not blinded. Skin measurements were not conducted under standardized conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No